CLINICAL TRIAL: NCT04797377
Title: Effects of Autologous Intraovarian Platelet Rich Plasma in Women With Poor Ovarian Response
Brief Title: Autologous Intraovarian Platelet Rich Plasma Treatment in Women With Poor Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 022019
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Poor Ovarian Reserve
Keywords: Platelet-Rich Plasma; Poor Ovarian Reserve; Oocyte Quality; Embryo Quality

STUDY DESIGN:
Intervention Model Description: After the women are recruited for the study, Antral follicle count (AFC), serum anti-mullerian hormone (AMH) and follicle stimulating hormone (FSH) levels will be determined at baseline and will be repeated beginning with the first menstrual cycle after treatment. Approximately 22 ml of blood sample will be collected under sterile conditions, and PRP will be prepared. The same day, within 1 hour of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into both ovaries. Ovarian reserve (AFC, FSH, AMH), and ICSI outcome parameters (number of MII oocytes, fertilization rate, oocyte and embryo quality) will be followed up to three months after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian Reserve (Experimental): Patients with diminished ovarian reserve or premature ovarian insufficiency
  Interventions: Biological: Autologous ovarian PRP injection

INTERVENTIONS:
Biological: Autologous ovarian PRP injection — The same day, within 1 hour of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into both ovaries using 11.8 inch (30 cm) single lumen 21G needles. The ovaries will be reached using needle guide preventing vascular or other structures rupture. The needle will be advanced into the centre of the ovarian medula without rotation. The correct tip placement will be confirmed by ultrasound. The activated PRP will be slowly introduced during careful retraction of the needle across the previously traversed ovarian cortex. The final PRP volume will be deposited under the ovarian capsule and the needle exit the ovary. Approximately 0.5 ml of the PRP solution will be injected into each ovary. After the procedure, the patients will be taken to the recovery room and will be observed for 30 minutes and also be discharged home on the same day.

SUMMARY:
Reproductive age women diagnosed with poor ovarian response (POR) based on Bologna criteria with a history of at least two prior failed ICSI cycle will be recruited for the study. Antral follicle count (AFC), serum anti-mullerian hormone (AMH), and early follicular phase serum follicle stimulating hormone (FSH) levels will determined at baseline. Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols and will be injected to both ovaries. Ovarian reserve parameters and ICSI outcomes will be determined.

DETAILED DESCRIPTION:
Reproductive age women diagnosed with POR based on Bologna criteria with a history of at least two prior failed intracytoplasmic sperm injection (ICSI) cycle will recruited for the study. Antral follicle count (AFC), serum anti-mullerian hormone (AMH), and early follicular phase serum follicle stimulating hormone (FSH) levels will be determined at baseline. Autologous blood obtained from peripheral vein will be used to prepare PRP following standard protocols. PRP injection will be performed under sedation anesthesia, using a 11.8 inch (30 cm) single lumen 21G needles under transvaginal ultrasound guidance. On the 2 to 4th days of the first three menstrual cycles following the procedure, AFC, AMH, and FSH levels will be re-assessed. Patients with at least one antral follicle will be started on ovarian stimulation for ICSI, followed by embryo transfer. Biomarkers of ovarian reserve (AFC, FSH, AMH), and ICSI outcome parameters (number of metaphase II (MII) oocytes, blastocyst embryos, fertilization rate, oocyte and embryo quality) will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with POR based on Bologna criteria and with a history of at least two prior failed ICSI cycles
* A previous assisted reproductive technology cycle with less than 3 oocytes (conventional stimulation protocol) and AFC < 7
* The same ovarian stimulation protocol before and after the PRP treatment

Exclusion Criteria:

* Age over 46 years,
* Body mass index (BMI) ≥ 30 kg/m2,
* Presence of pregnancy
* Uncontrolled endocrine disorders (polycystic ovary syndrome and others)
* Parental genetic and chromosomal disorders,
* Immunological disorders
* Cancer diagnostics

Ages: 30 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Based on gender identity
Enrollment: 66 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Oocyte number | 3 months
  Number of Metaphase II oocyte yield.
Oocyte quality | 3 months
  Oocytes will be classified based on morphological assessment and enumeration of extracytoplasmic anomalies.
Embryo number | 3 months
  Number of produced embryos per cycle.
Embryo quality | 3 months
  Morphological evaluation of the cultured embryos will be conducted 120 or 144 hr following sperm injection. Blastocysts scoring will be performed on day 5 or 6 depending on the blastocoel cavity expansion and on the inner cell mass and trophectoderm cells integrity.
Fertilization rate | 3 months
  Fertilization rate will be calculated as the percentage of transformation of the injected oocytes into two pronuclei.

SECONDARY OUTCOMES:
Antral follicle count (AFC) | 3 months
  Number of Antral Follicles determined by pelvic sonogram on day 2 or 3 of the cycle.
Serum anti-mullerian hormone (AMH) | 3 months
  Serum concentration of anti-mullerian hormone determined on day 3 of the cycle by an electrochemiluminescent (ECLIA) immunoanalyzer.
Serum follicle stimulating hormone (FSH) | 3 months
  Serum concentration of follicle stimulating hormone (FSH) levels determined on day 3 of the cycle by an electrochemiluminescent (ECLIA) immunoanalyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Nadezhda Women's Health Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drakopoulos P, Bardhi E, Boudry L, Vaiarelli A, Makrigiannakis A, Esteves SC, Tournaye H, Blockeel C. Update on the management of poor ovarian response in IVF: the shift from Bologna criteria to the Poseidon concept. Ther Adv Reprod Health. 2020 Jul 31;14:2633494120941480. doi: 10.1177/2633494120941480. eCollection 2020 Jan-Dec. PMID 32844159
- [Background] Zhang Y, Zhang C, Shu J, Guo J, Chang HM, Leung PCK, Sheng JZ, Huang H. Adjuvant treatment strategies in ovarian stimulation for poor responders undergoing IVF: a systematic review and network meta-analysis. Hum Reprod Update. 2020 Feb 28;26(2):247-263. doi: 10.1093/humupd/dmz046. PMID 32045470
- [Background] Panda SR, Sachan S, Hota S. A Systematic Review Evaluating the Efficacy of Intra-Ovarian Infusion of Autologous Platelet-Rich Plasma in Patients With Poor Ovarian Reserve or Ovarian Insufficiency. Cureus. 2020 Dec 12;12(12):e12037. doi: 10.7759/cureus.12037. PMID 33457137
- [Background] Everts P, Onishi K, Jayaram P, Lana JF, Mautner K. Platelet-Rich Plasma: New Performance Understandings and Therapeutic Considerations in 2020. Int J Mol Sci. 2020 Oct 21;21(20):7794. doi: 10.3390/ijms21207794. PMID 33096812
- [Background] Sills ES, Wood SH. Autologous activated platelet-rich plasma injection into adult human ovary tissue: molecular mechanism, analysis, and discussion of reproductive response. Biosci Rep. 2019 Jun 4;39(6):BSR20190805. doi: 10.1042/BSR20190805. Print 2019 Jun 28. PMID 31092698
- [Background] Bos-Mikich A, de Oliveira R, Frantz N. Platelet-rich plasma therapy and reproductive medicine. J Assist Reprod Genet. 2018 May;35(5):753-756. doi: 10.1007/s10815-018-1159-8. Epub 2018 Mar 21. PMID 29564738
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008